CLINICAL TRIAL: NCT05155332
Title: Phase I Open-label, Dose Escalation Trial of BI 1831169 Monotherapy and in Combination With an Anti-PD-1 mAb in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Study to Test Different Doses of BI 1831169 Alone and in Combination With an Anti-PD-1 Antibody in People With Different Types of Advanced Cancer (Solid Tumors)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1456-0001; 2020-003902-30 (EudraCT Number)
Record Dates: First submitted 2021-12-10; First posted 2021-12-13 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors
MeSH Terms: interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1 (Monotherapy): Arm A (Experimental)
  Interventions: Drug: BI 1831169
- Part 1 (Monotherapy): Arm B (Experimental)
  Interventions: Drug: BI 1831169
- Part 1 (Monotherapy): Arm C (Experimental)
  Interventions: Drug: BI 1831169
- Part 2 (Combination therapy): Arm D (Experimental)
  Interventions: Drug: BI 1831169; Drug: anti-PD-1 antibody
- Part 2 (Combination therapy): Arm E (Experimental)
  Interventions: Drug: BI 1831169; Drug: anti-PD-1 antibody
- Part 2 (Combination therapy): Arm F (Experimental)
  Interventions: Drug: BI 1831169; Drug: anti-PD-1 antibody
- Part 2 (Combination therapy): Arm G (Experimental)
  Interventions: Drug: BI 1831169; Drug: anti-PD-1 antibody

INTERVENTIONS:
Drug: BI 1831169 — BI 1831169
Drug: anti-PD-1 antibody — anti-PD-1 antibody
  Arms: Part 2 (Combination therapy): Arm D; Part 2 (Combination therapy): Arm E; Part 2 (Combination therapy): Arm F; Part 2 (Combination therapy): Arm G

SUMMARY:
This study is open to adults with different types of advanced cancer (solid tumors) that are accessible for injection and/or biopsy. This is a study for people with a life expectancy of at least 3 months after starting study treatment. The purpose of this study is to find the highest dose of a medicine called BI 1831169 that people with advanced cancer can tolerate when taken with or without a type of antibody called a checkpoint inhibitor (anti-PD-1 antibody). Another purpose is to check whether the study treatment can fight cancer. In this study, BI 1831169 is given to people for the first time.

This study has 2 parts. In Part 1, participants get BI 1831169 alone for up to 3 months. In Part 2, participants get BI 1831169 in combination with a checkpoint inhibitor. Participants who take the combination treatment get BI 1831169 for up to 3 months and a checkpoint inhibitor for up to 1 year. BI 1831169 is given as an injection into the tumor, or as an infusion into the vein, or both (injection and infusion). Checkpoint inhibitors are given as an infusion into a vein. Participants get the medicines about every 3 weeks. This is called a treatment cycle.

Participants visit the site study site regularly. The number of study visits vary based on the study phase and treatment response. Some visits include an overnight stay. The doctors regularly check the participants' health and monitor the tumors. The doctors also take note of any health problems that could have been caused by the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced, unresectable and/or metastatic or relapsed/refractory solid tumors
* At least one or two accessible lesions, one with a minimum lesion diameter for injection of BI 1831169 (where applicable), and one which is amenable to biopsy (where applicable). Lesions must either be easily accessible or, if not easily accessible, patient must be willing to undergo repeated procedures (e.g., image guided procedures) for both biopsies and injections of BI 1831169
* Has failed conventional treatment or for whom no therapy of proven efficacy exists, who is not eligible for established treatment options. Patient must have exhausted available treatment options known to prolong survival for their disease. This criterion does not apply to the specific indications in Part 2.

Further inclusion criteria apply.

Exclusion Criteria:

* Previous treatment with Vesicular stomatitis virus (VSV)-based agents
* Concomitant medication or condition considered a high risk for complications from injection or biopsy as per the Investigator's judgement
* Presence of brain metastases
* Presence of Human Immunodeficiency Virus (HIV) meeting certain criteria, active autoimmune disease or chronic active infection (Hepatitis C or B virus (HCV/HBV))
* Chronic steroid use, regardless of daily dose Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2027-12-13 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Part 1.1, Dose escalation/Confirmation: Occurrence of Dose limiting toxicities (DLTs) during the mono Maximum tolerated dose (MTD) evaluation period | up to 21 days
  Part 1 (Monotherapy).
Part 1.2, Dose expansion: Objective response (OR) defined as best overall response (BOR) of confirmed intratumoral immunotherapy complete response (itCR) or confirmed intratumoral immunotherapy partial response (itPR) | up to 49 months
  BOR is defined according to Response Criteria for Intratumoral Immunotherapy in Solid Tumors (itRECIST).
  BOR will consider all tumor assessments from first administration of trial medication until disease progression or death (whichever occurs first) or last evaluable tumor assessment before start of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent.
Part 2.1, Dose escalation/Confirmation: Occurrence of Dose limiting toxicities (DLTs) during the combination Maximum tolerated dose (MTD) evaluation period | up to 21 days
  Part 2 (Combination Therapy).
Part 2.2, Dose Expansion, Arm D: Objective response (OR) defined as best overall response (BOR) of confirmed intratumoral immunotherapy complete response (itCR) or confirmed intratumoral immunotherapy partial response (itPR) | up to 49 months
  BOR is defined according to Response Criteria for Intratumoral Immunotherapy in Solid Tumors (itRECIST).
  BOR will consider all tumor assessments from first administration of trial medication until disease progression or death (whichever occurs first) or last evaluable tumor assessment before start of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent.
Part 2.2, Dose Expansion, Arm E, Arm F, Arm G: Objective response (OR) defined as best overall response (BOR) of confirmed immunotherapy complete response (iCR) or confirmed immunotherapy partial response (iPR) | up to 49 months
  BOR is defined according to Response Criteria for intravenous Immunotherapy in Solid Tumors (iRECIST).
  BOR will consider all tumor assessments from first administration of trial medication until disease progression or death (whichever occurs first) or last evaluable tumor assessment before start of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent.

SECONDARY OUTCOMES:
Part 1.1, Dose escalation/Confirmation: Occurrence of DLTs during the on-treatment period | up to 49 months
Part 1.1, Dose escalation/Confirmation: Occurrence of adverse events during the on-treatment period | up to 49 months
Part 1.2, Dose expansion: Occurrence of adverse events during the on-treatment period | up to 49 months
Part 1.2, Dose expansion: Occurrence of DLTs during the mono MTD evaluation period | up to 49 months
Part 2.1, Dose escalation/Confirmation: Occurrence of DLTs during the on-treatment period | up to 49 months
Part 2.1, Dose escalation/Confirmation: Occurrence of adverse events during the on-treatment period | up to 49 months
Part 2.2 - Dose Expansion by Indication, All Arms: Occurrence of adverse events during the on-treatment period | up to 49 months
Part 2.2 - Dose Expansion by Indication, Arm D: Duration of objective response (DoR) | up to 49 months
  DoR is defined as the time from first documented itCR or itPR according to modified itRECIST until the earliest of disease progression or death among patients with OR.
Part 2.2, Dose Expansion by Indication, Arm D: Disease control (DC) | up to 49 months
  DC is defined as a BOR itCR, itPR or intratumoral immunotherapy stable disease (itSD), with BOR defined according to modified itRECIST.
Part 2.2, Dose Expansion by Indication, Arms E, F, G: Duration of objective response (DoR) | up to 49 months
  DoR is defined as the time from first documented iCR or iPR according to iRECIST until the earliest of disease progression or death among patients with OR.
Part 2.2, Dose Expansion by Indication, Arms E, F, G: Disease control (DC) | up to 49 months
  DC is defined as a BOR of iCR, iPR or immunotherapy stable disease (iSD), with BOR defined according to iRECIST.
Part 2.2, Dose Expansion by Indication, Arm E: Progression-Free Survival (PFS) rate at 4 months | up to 4 months
  PFS rate at 4 months (PFS-4) according to iRECIST is defined as the proportion of patients who are alive and without progression by 4 months from the start of treatment.

CONTACTS AND LOCATIONS:
Locations (40):
- United States (14):
  - Banner MD Anderson Cancer Center-Gilbert-55251, Gilbert, Arizona
  - University of Arizona, Tucson, Arizona
  - University of California San Diego, La Jolla, California
  - Providence St. John's Health Center, Santa Monica, California
  - University of Colorado Denver, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - University of Louisville, Louisville, Kentucky
  - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - Morristown Medical Center, Morristown, New Jersey
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Prisma Health, Greenville, South Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Southern Oncology Clinical Research Unit, Bedford Park, South Australia
  - Peninsula Haematology & Oncology, Frankston, Victoria
- Austria (2):
  - Medical University of Innsbruck, Innsbruck
  - Salzburg Cancer Research Institute, Salzburg
- Belgium (3):
  - Edegem - UNIV UZ Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven, Leuven
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- France (4):
  - INS Bergonie, Bordeaux
  - HOP Timone, Marseille
  - CTR Eugène Marquis, Rennes
  - INS Gustave Roussy, Villejuif
- Germany (4):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Italy (3):
  - Istituto Di Candiolo, Candiolo (TO)
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Spain (5):
  - Hospital Quiron. I.C.U., Barcelona
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Fundación Jiménez Díaz, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Instituto Valenciano de Oncología, Valencia
- Switzerland (2):
  - University Hospital Bern, Bern
  - University Hospital Geneva, Geneva

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Porosnicu M, Quinson AM, Crossley K, Luecke S, Lauer UM. Phase I study of VSV-GP (BI 1831169) as monotherapy or combined with ezabenlimab in advanced and refractory solid tumors. Future Oncol. 2022 Aug;18(24):2627-2638. doi: 10.2217/fon-2022-0439. Epub 2022 Jun 14. PMID 35699077
- See also: Related Info — https://www.mystudywindow.com